CLINICAL TRIAL: NCT01421693
Title: Randomized, Open-label, Superiority Trial of the Effectiveness of Gatifloxacin Versus Ceftriaxone for the Treatment of Uncomplicated Enteric Fever.
Brief Title: Gatifloxacin Versus Ceftriaxone in the Treatment of Enteric Fever
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: University of Oxford (Other); Patan Academy of Health Sciences, Nepal (Unknown); Patan Hospital, Nepal (Unknown); Civil Hospital, Nepal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03NP
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Enteric Fever; Typhoid Fever
Keywords: Gatifloxacin; Ceftriaxone; Enteric fever; Typhoid fever
MeSH Terms: conditions — Typhoid Fever | interventions — Ceftriaxone; Gatifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gatifloxacin (Active Comparator): Gatifloxacin 10mg/kg/day for 7 days
  Interventions: Drug: Gatifloxacin
- Ceftriaxone (Active Comparator): * ≥2-<14 years - 60mg/kg/ once daily for 7 days
  * 14 years and older - 2g once daily for 7 days
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Ceftriaxone — * ≥2-<14 years - 60mg/kg/ once daily for 7 days
  * 14 years and older - 2g once daily for 7 days
  * Intravenous infusion. Vials of crystalline powder.
  Arms: Ceftriaxone
Drug: Gatifloxacin — Gatifloxacin 10 mg/kg/day for 7 days. Tablets for oral administration.
  Arms: Gatifloxacin

SUMMARY:
The investigators aim to compare two antibiotic treatments for enteric (typhoid) fever. Three hundred patients at Patan Hospital will be enrolled in the study. Patients will be assigned to one of the two treatments by chance and followed for 6 months. The two treatment groups will be compared to see which treatment is more likely to make the patient better.

DETAILED DESCRIPTION:
With the study hypothesis that Gatifloxacin is superior to Ceftriaxone in terms of treatment failure in patients with enteric fever, a comparative study will be conducted at Patan Hospital. 300 patients who are diagnosed with enteric fever will be enrolled into the study. The patients will be randomized to one of two groups. One group will receive treatment with Gatifloxacin for 7 days, and the other with Ceftriaxone. The patients will be followed during the treatment courses and at several points of 6 months after initial presentation. The endpoints then will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or culture proven enteric fever
* >= 2 <= 45 years of age
* Fever >= 38°C for >= 4 days
* Informed consent to participate in the study

Exclusion Criteria:

* Pregnancy
* Obtundation
* Shock
* Visible jaundice
* Presence of signs of gastrointestinal bleeding
* Evidence of severe disease
* Diabetes
* History of hypersensitivity to either of the trial drugs
* Known previous treatment with a quinolone antibiotic or 3rd generation cephalosporin or macrolide within one week of hospital admission.

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Rate of treatment failure | upon occurance, within 28 days
  Any one (1) of the following defines treatment failure:
  * Fever clearance time >7 x 24hours post treatment initiation
  * Blood culture positive at Day 8 of treatment (microbiological failure)
  * Requirement of rescue treatment
  * Culture confirmed or syndromic relapse within 28 days of initiation of treatment
  * The development on treatment of any enteric fever related complication within 28 days of initiation of treatment including, clinically significant bleeding, fall in the Glasgow Coma Score, perforation of the gastrointestinal tract or admission to hospital Both the absolute risk of treatment failure and the time to treatment failure will be analyzed

SECONDARY OUTCOMES:
S.typhi or S.paratyphi carriage | 1 month, 3 months and 6 months
  Stool culture positive for S.typhi or S.paratyphi carriage
Number of adverse events | within 6 months
  Treatment tolerance as defined by the number of adverse events, serious adverse events and disease complications
Household transmission | within 6 months
  Total number of febrile episodes, hospital visits and hospital admissions within household members
Time to fever clearance | upon occurance, within 7 days
  Time from first dose of treatment until a temperature which is ≤37•5°C for a 48 hour period is first recorded.
Rate of culture-positive and syndromic clinical relapses | within 28 days of starting therapy
Rate of relapses confirmed using additional diagnostic techniques | within 28 days of starting therapy
  Additional techniques will include culture-PCR and gene expression profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Buddha Basnyat, MD, Principal Investigator — University of Oxford
Locations (2):
- Nepal (2):
  - Civil Hospital, Kathmandu
  - Patan Hospital, Kathmandu

REFERENCES:
- [Derived] Arjyal A, Basnyat B, Nhan HT, Koirala S, Giri A, Joshi N, Shakya M, Pathak KR, Mahat SP, Prajapati SP, Adhikari N, Thapa R, Merson L, Gajurel D, Lamsal K, Lamsal D, Yadav BK, Shah G, Shrestha P, Dongol S, Karkey A, Thompson CN, Thieu NTV, Thanh DP, Baker S, Thwaites GE, Wolbers M, Dolecek C. Gatifloxacin versus ceftriaxone for uncomplicated enteric fever in Nepal: an open-label, two-centre, randomised controlled trial. Lancet Infect Dis. 2016 May;16(5):535-545. doi: 10.1016/S1473-3099(15)00530-7. Epub 2016 Jan 20. PMID 26809813
- See also: Oxford University Clinical Research Unit, Viet Nam — http://www.oucru.org
- See also: Oxford University Clinical Research Unit, Nepal — http://www.tropicalmedicine.ox.ac.uk/nepal
- See also: Trial Ethical Approval letters and Informed Consent Forms — http://www.oucru.org/index.php?option=com_content&view=article&id=336&Itemid=111&lang=en